CLINICAL TRIAL: NCT01373554
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, A Multicenter, Randomized, Double-blind, Placebo-controlled, 3 Parallel Groups, Phase 2 Study to Evaluate the Efficacy, Safety and Pharmacokinetics of Oltipraz in Patients With Non-alcoholic Fatty Liver Disease (Except Liver Cirrhosis)
Brief Title: Efficacy and Safety of Oltipraz in the Patients With Non-alcoholic Fatty Liver Disease
Acronym: PMK-N01GI1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PharmaKing (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PMK-N01GI1
Record Dates: First submitted 2011-06-03; First posted 2011-06-15 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Non-alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — oltipraz

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Oltipraz (Experimental)
  Interventions: Drug: Oltipraz

INTERVENTIONS:
Drug: Placebo — 30mig/bid or 60mg/bid P.O
  Arms: Placebo
Drug: Oltipraz — 30mig/bid or 60mg/bid P.O
  Arms: Oltipraz

SUMMARY:
Dithiolethiones, a novel class of adenosine monophosphate-activated protein kinase (AMPK) activators, prevent insulin resistance through AMPK-dependent p70 ribosomal S6 kinase-1 (S6K1) inhibition. And it is well known that the modulation of S6K1 by oltipraz inhibited the development of insulin resistance and hyperglycemia through the AMPK-S6K1 pathway.Also some research reported that LXRg (a member of the nuclear hormone receptor)-mediated increases in SREBP-1c (the sterol regulatory element-binding protein-1c gene) promote the expression of lipogenic genes and enhance fatty acid synthesis and oltipraz inhibits LXRg and SREBP-c. Therefore, Oltipraz inhibits fatty acid synthesis through AMPK-S6K1 pathway and LXRg-SREBP-1c pathway in liver.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18, under 75 years of age
* Patients with non-alcoholic fatty liver disease

Exclusion Criteria:

* Over 2 ratio of AST to ALT
* Type 1 diabetes mellitus (insulin-dependent diabetes mellitus)
* Disorder in liver function with an exception of non-alcoholic fatty liver (e.g. Virus infection, biliary atresia, autoimmune hepatitis and etc.)
* Patients who have been taken drugs induced fatty liver for over 3 month within 1 year of participation in this study; amiodarone, tamoxifen, methotrexate, tetracyclines, glucocorticoids, anabolic steroids, over usual dose of estrogen for hormone replacement therapy and valproate
* Patients who has been taken any medications that could affect the treatment for non-alcoholic steatohepatitis: insulin, insulin sensitizer(metformin, thiazolidinedione), high dose of vitamin E, high dose of UDCA, pentoxifylline, SAM-e, Betaine, types of Statin, types of fibrate and orlistat
* Patients who had a Bariatric surgery less than 6 month prior to the participation in the study
* Patients who are judged by investigator that participation of the study is difficult due to disease as follow; hepatic cirrhosis, Wilson's disease, malignant tumor, serious metabolic disease, severe renal disease, severe pulmonary disease, severe cardiovascular disease, severe nervous disease/psychiatric disorder, muscle disease and etc
* Any history of immune disorder which affect the changes in cytokine:

inflammatory bowel disease, autoimmune thrombocytopenic purpura, system lupus erythematosus, autoimmune hemolytic anemia, severe psoriasis, rheumatic arthritis and etc

* Patients who have received treatment that may affect liver function within 1 month prior to the participation in the study
* Patient who has been administered other investigational product within 1 month prior to the participation in the study
* Patient who is not allowed to get MRS test: pacemaker, shunt and etc
* Pregnant or nursing women
* Patient who considered ineligible for participation in the study as Investigator's judgment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-05; Primary Completion 2013-06 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
MRS | 24 weeks
  To evaluate the efficacy of the Oltipraz on change in quantity of liver fat concentration assessed by MRS from baseline to 24 weeks in patients with non-alcoholic fatty liver disease

SECONDARY OUTCOMES:
change in ALT, AST and total bilirubin | 24 weeks
change in Cholesterol, Triglyceride | 24 weeks
change in HOMA-IR | 24 weeks
change in BMI | 24 weeks
changes in NAS | 24 weeks
  Subjects with liver biopsy:

CONTACTS AND LOCATIONS:
Overall Officials: YoonJun Kim, MD.PhD, Principal Investigator — Seoul National University Hospital
Locations (5):
- South Korea (5):
  - Inje University Ilsan Paik Hospital, Dahwa-dong, Ilsanseo-gu, Goyang-si, Gyeonggi-do
  - NHUS Ilsan Hospital, Ilsan-ro Ilsan-donggu, Goyang-si
  - Seoul National University Hospital, Daehak-ro Jongno-gu, Seoul
  - Korea University Guro hospital, Gurodong-ro, Seoul
  - Boramae Hospital, Sindaebang-dong Dongjak-gu, Seoul

REFERENCES:
- [Background] Kim SG, Kim YM, Choi YH, Lee MG, Choi JY, Han JY, Cho SH, Jang JW, Um SH, Chon CY, Lee DH, Jang JJ, Yu ES, Lee YS. Pharmacokinetics of oltipraz and its major metabolite (RM) in patients with liver fibrosis or cirrhosis: relationship with suppression of circulating TGF-beta1. Clin Pharmacol Ther. 2010 Sep;88(3):360-8. doi: 10.1038/clpt.2010.89. Epub 2010 Jul 21. PMID 20664537
- [Derived] Kim W, Kim BG, Lee JS, Lee CK, Yeon JE, Chang MS, Kim JH, Kim H, Yi S, Lee J, Cho JY, Kim SG, Lee JH, Kim YJ. Randomised clinical trial: the efficacy and safety of oltipraz, a liver X receptor alpha-inhibitory dithiolethione in patients with non-alcoholic fatty liver disease. Aliment Pharmacol Ther. 2017 Apr;45(8):1073-1083. doi: 10.1111/apt.13981. Epub 2017 Feb 22. PMID 28225186
- See also: Oltipraz — http://druginfo.nlm.nih.gov/drugportal/ProxyServlet?mergeData=true&objectHandle=DBMaint&APPLICATION_NAME=drugportal&actionHandle=default&nextPage=jsp/drugportal/ResultScreen.jsp&TXTSUPERLISTID=0064224211&QV1=OLTIPRAZ